CLINICAL TRIAL: NCT00369694
Title: Randomized Double Blind Dummy Controlled Trial Of 24 Versus 72 Hours Of Terlipressin As An Adjuvant Therapy In Acute Variceal Bleed
Brief Title: Short Course Terlipressin for Control of Acute Variceal Bleeding
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Aga Khan University (Other)
Collaborators: Ferozsons Laboratories Ltd. (Industry)
Responsible Party: Ethical Review Committee (ERC), The Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 446-Med/ERC-05
Record Dates: First submitted 2006-08-24; First posted 2006-08-29 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Hemorrhage; Esophageal Varices; Portal Hypertension
Keywords: Esophageal varices; Portal Hypertension; Melena; Hematemesis; Gastrointestinal Hemorrhage; Terlipressin; Efficacy; Safety
MeSH Terms: conditions — Hemorrhage; Esophageal and Gastric Varices; Hypertension, Portal; Melena; Hematemesis; Gastrointestinal Hemorrhage | interventions — Terlipressin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): 72 hours of Terlipressin
  Interventions: Drug: Terlipressin
- 2 (Placebo Comparator): 24 hours of Terlipressin & then next 48 hours of Dummy of Terlipressin
  Interventions: Drug: Terlipressin & then Dummy

INTERVENTIONS:
Drug: Terlipressin — 2 mg Terlipressin stat, then 1 mg q6h for total of 72 hours
  Other Names: Novapressin
  Arms: 1
Drug: Terlipressin & then Dummy — 2 mg Terlipressin stat then 1 mg q6 hours for 24 hours, then a Dummy of Terlipressin q6 hours for the next 48 hours.
  Other Names: Novapressin
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether 24 hours of Terlipressin is as effective as 72 hours of Terlipressin in preventing re-bleed once esophageal variceal bleed has been controlled with endoscopic therapy (variceal band ligation or sclerotherapy) in low to moderate risk variceal bleed patients and hence can save cost and may decrease length of hospital stay especially in the I.C.U or high dependency units.

DETAILED DESCRIPTION:
The esophageal variceal bleeding is usually controlled with endoscopic treatment of variceal band ligation or sclerotherapy along with vasoactive drugs like Terlipressin or Octreotide. The risk of re-bleeding is highest during the initial 5 days from first presentation. Terlipressin is usually given for 3 days (72 hours). In this study we are trying to prove that among low to moderate risk patients, a short course of 1 day (24 hours) of Terlipressin is as effective as 3 days (72 hours) in preventing re-bleed once bleeding has been controlled with endoscopic therapy. This intervention will save 2 days cost incurred on the Terlipressin and may also help in decreasing the length of hospital stay in future.

ELIGIBILITY:
Inclusion Criteria:

* Acute esophageal variceal bleed
* Liver cirrhosis
* Child's score </= 11

Exclusion Criteria:

* Patient on Mechanical ventilator and or ionotropic support
* Active angina, Recent Myocardial infarction or dynamic EKG changes
* Failure to control variceal bleed on initial endoscopy
* Gastric variceal bleed
* Spontaneous bacterial peritonitis at presentation
* Hepatocellular carcinoma or other liver metastatic malignancy
* Portal vein thrombosis

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-08; Primary Completion 2008-07 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Variceal Re-bleed | 120 hours (5 Days)

SECONDARY OUTCOMES:
All cause 30 days mortality | 30 days
30 days rebleed | 30 days from index bleed
Safety of Terlipressin | In Hospital safety

CONTACTS AND LOCATIONS:
Overall Officials: Saeed S Hamid, FRCP, FACG, Study Chair — The Aga Khan University Hospital; Zahid SM Azam, MBBS, FCPS, Study Director — The Aga Khan University Hospital; Wasim SM Jafri, FRCP, FACG, Study Director — The Aga Khan University Hospital
Locations (1):
- The Aga Khan University Hospital, Karachi, Sindh, Pakistan